CLINICAL TRIAL: NCT07136805
Title: A Multi-center, Randomized, Single-masked, Active-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of 1.0% VVN461 Ophthalmic Solution in Patients With Non-infectious Anterior Uveitis
Brief Title: A Phase 3 Study of VVN461 Ophthalmic Solution for Noninfectious Anterior Uveitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VivaVision Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VVN461-CCS-301
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Non-infectious Anterior Uveitis
MeSH Terms: interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- VVN461, 1.0% (Experimental): VVN461 Ophthalmic Solution, 1.0%
  Interventions: Drug: VVN461 Ophthalmic Solution 1.0%
- 1.0% prednisolone acetate (Active Comparator): 1.0% prednisolone acetate, Pred Forte
  Interventions: Drug: 1.0% prednisolone acetate

INTERVENTIONS:
Drug: VVN461 Ophthalmic Solution 1.0% — 1 drop for study eye each time, 6 times daily (Q2h) for 7 days; 4 times daily (QID) for 7 days; 2 times daily (BID) for 7 days; 1 time daily for 7 days
  Arms: VVN461, 1.0%
Drug: 1.0% prednisolone acetate — 1 drop for study eye each time, 6 times daily (Q2h) for 7 days; 4 times daily (QID) for 7 days; 2 times daily (BID) for 7 days; 1 time daily for 7 days
  Arms: 1.0% prednisolone acetate

SUMMARY:
This is a multicenter, randomized, single-masked, active-controlled, parallel, Phase III pivotal study in China

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent form (ICF), the subject must be aged 18 to 70 years (inclusive);
* At screening, the affected eye is diagnosed with non-infectious anterior uveitis (acute or recurrent acute, only unilateral eye affected patients are included);
* At screening, the ACC grade of the affected eye is 2+ or 3+ [SUN criteria];
* At screening, the ACF grade of the affected eye is ≥1 [SUN criteria];

Exclusion Criteria:

* At screening, the affected eye has an ACC grade of 4+ or hypopyon
* Diagnosis of intermediate uveitis, posterior uveitis, or panuveitis in either eye at the time of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in anterior chamber cell (ACC) grade in the study eye at Day 14 | Day 14

SECONDARY OUTCOMES:
The proportion of subjects with ACC grade of 0 in the study eye at Day 14 | Day 14

IPD SHARING:
Plan to Share IPD: No